CLINICAL TRIAL: NCT04460131
Title: Association Between Soluble ST2 and Cardiovascular Outcome After Cardiovascular Surgery
Brief Title: Soluble ST2 and Cardiovascular Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Nanjing Medical University, Nanjing Medical University
Other Study IDs: sST2-2019
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: soluble ST2 — Serum sST2 was measured on a monoclonal electrochemiluminescence immunoassay. Samples were exposed to two freeze cycles before analysed. Samples were exposed to two thawfreeze cycles before analysed.

SUMMARY:
Cardiac surgery induces hemodynamic stress on the myocardium, and this process can be associated with significant cardiovascular morbidity and mortality. Soluble suppression of tumorigenicity 2 (sST2) is biomarker of myocardial remodeling and fibrosis; however, little is known regarding their potential association with cardiovascular events. This study aimed to investigate the release of sST2 and its association with cardiovascular events undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Congenital heart disease requiring surgery
* Valvular heart disease requiring surgery
* Arrhythmia requiring surgery
* Aortic dissection requiring surgery
* Coronary heart disease requiring surgery

Exclusion Criteria:

* age <18 years
* pregnancy
* severe renal dysfunction (creatinine >200µmol/L)
* not capable of understanding or signing informed consent.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adults patients with heart disease who underwent cardiac surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days after surgery
  Number of participants death of 30 days after surgery

SECONDARY OUTCOMES:
Heart failure | 30 days after surgery
  requiring initiation or change in heart failure medication or requiring hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China